CLINICAL TRIAL: NCT06524505
Title: Efficacy, Tolerability, and Cognitive Effects of Deep Transcranial Magnetic Stimulation for Bipolar Depression: a Double-blind, Randomized Controlled Trial
Brief Title: Efficacy, Tolerability, and Cognitive Effects of Deep Transcranial Magnetic Stimulation for Bipolar Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dTMS-TJAH
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-05

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dTMS group (Experimental): Participants receive active stimulation with H1 coil, consisting of 55 18 Hz, 2 s trains at 120% MT intensity, with a between-train interval of 20 s ,1980 pulses per day. The subjects were stimulated every day for 4 weeks (except weekends).
  Interventions: Device: deep Transcranial Magnetic Stimulation (dTMS) -active
- sham group (Sham Comparator): The sham stimulation was performed using the same procedures, with the sham coil.
  Interventions: Device: deep Transcranial Magnetic Stimulation (dTMS) -sham

INTERVENTIONS:
Device: deep Transcranial Magnetic Stimulation (dTMS) -active — with the H1-coil device included 20-min sessions of 18 Hz (2-s trains separated by 20-s inter-train intervals, 55 trains totaling 1980 pulses/session).
  Arms: dTMS group
Device: deep Transcranial Magnetic Stimulation (dTMS) -sham — The sham stimulation was performed using the same procedures, with the sham coil.
  Arms: sham group

SUMMARY:
The aim of this study is to evaluate the feasibility and efficacy of deep transcranial magnetic stimulation (dTMS) as an add-on treatment for bipolar depression. Meanwhile, we aim to evaluate the effect of dTMS on cognitive function of bipolar depressive patients. we hypothesize dTMS would improve depressive symptoms and cognitive function in bipolar disorder.

DETAILED DESCRIPTION:
This is a randomized, double-blind, sham-controlled study to detect the effect of dTMS for treatment of bipolar depression. 100 participants were randomly assigned 1:1 to dTMS group or sham-control group. For both active and sham group, daily dTMS sessions were scheduled in a 5-day sequence for four consecutive weeks, and each session lasted 20minutes. Based on the original and stable medication, the active stimulation consisted of 55 18 Hz, 2 s trains at 120% MT intensity, with a between-train interval of 20 s (1980 pulses per day or 39 600 pulses per treatment). The sham stimulation was performed using the same procedures, with the sham coil.

Scale assessments are performed at baseline, week 2, week 4 and week 8. Collection of blood took place at baseline, week 4 and week 8.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of bipolar depression;

* Met standardized criteria for failure to achieve remission from pharmacological treatment in the current illness episode;
* Pharmacological treatment maintained unchanged for the four weeks preceding rTMS application；
* Able to read, verbalize understanding and voluntarily sign the informed consent form prior to performance of any study-specific procedures or assessments

Exclusion Criteria:

* Previous treatment with rTMS;
* Ferromagnetic material close to the head;
* Cardiac pacemaker and/or implanted electronic device;
* The presence of neurological disorders (uncontrolled epilepsy, previous significant head injuries, brain surgery);
* Pregnancy or lactation;
* Significant medical and/or psychiatric comorbidities;
* Substance abuse in the last three months (not including caffeine or nicotine);
* Acute psychosis;
* Acute suicidality;
* Patient refuses to sign consent for participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
The change over time in the score of Hamilton Depression Rating Scale (HDRS-17). | baseline, week 2, week 4, week 8
  The aim is to explore whether dTMS combined with Pharmacological treatment could alleviate the severity of depressive symptoms as measured with HDRS-17 in bipolar depression after 4-week treatment. Hamilton Depression Rating Scale (HDRS-17) was used to evaluate the severity of symptoms of depression. Higher total score of the scale means more severe depressive symptoms.

SECONDARY OUTCOMES:
The change over time in the score of Hamilton Anxiety Rating Scale (HAMA) | baseline, week 2, week 4, week 8
  The aim is to explore whether dTMS combined with Pharmacological treatment could alleviate the severity of anxious symptoms as measured with HAMA in bipolar depression after 4-week treatment. Hamilton Anxiety Rating Scale (HAMA) was used to evaluate the severity of symptoms of anxiety. Higher total score of the scale means more severe anxious symptoms.
The change of scores in MATRICS Consensus Cognitive Battery(MCCB) | baseline, week 4, week 8
  The aim is to observe whether active-stimuli in addition to pharmacological treatment will improve the cognitive function as measured with the MATRICS Consensus Cognitive Battery (MCCB) after 4 weeks of treatment compared to sham-stimuli, and investigators assess the scale at baseline, week 4 and week 8.
The changes of levels of Brain Derived Neurotrophic Factor in peripheral blood | baseline, week 4, week 8
  The aim is to investigate the change of Brain Derived Neurotrophic Factor level in peripheral blood as active stimuli in addition to regular medical treatment after 4 weeks of treatment compared to sham stimuli, and EDTA tubes were used to collect 5ml of peripheral blood at baseline, weeks 4, and 8 before feeding. The plasma was extracted after centrifugation, and the concentration of BDNF in plasma was detected by ELISA.
The change of scores of Adverse events scale from baseline to week 4 | baseline, week 4
  The aim is to evaluate the adverse effects during the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, China